CLINICAL TRIAL: NCT01026636
Title: An Open-Label Study to Evaluate the Single-Dose Pharmacokinetics and Safety of Ceftobiprole in Pediatric Patients =3 Months to 17<18 Years of Age, Undergoing Treatment With Systemic Antibiotics
Brief Title: A Single-Dose Pharmacokinetics and Safety Study of Ceftobiprole in Pediatric Patients =3 Months to <18 Years of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CR012304; CSI-1001 (Other: Basilea)
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Staphylococcal Skin Infections; Streptococcal Infections
Keywords: Staphylococcal Skin Infections; Skin Infections; Streptococcal Infections
MeSH Terms: conditions — Staphylococcal Skin Infections; Streptococcal Infections; Cellulitis | interventions — ceftobiprole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ceftobiprole (Experimental): Ceftobiprole 7mg/kg - 15mg/kg per day as 2h infusion
  Interventions: Drug: Ceftobiprole

INTERVENTIONS:
Drug: Ceftobiprole
  Other Names: Ceftobiprole 7mg/kg - 15kg/kg per day as 2h infusion

SUMMARY:
This study will assess the pharmacokinetics (how drugs are absorbed, distributed in the body and removed over time) and safety of a single dose of ceftobiprole in pediatric patients undergoing treatment with systemic antibiotics and may be used to guide dosing recommendations for ceftobiprole in children.

DETAILED DESCRIPTION:
This purpose of this study will be to assess the pharmacokinetics (how drugs are absorbed, distributed in the body and removed over time) and safety of a single dose of ceftobiprole in pediatric patients undergoing treatment with systemic antibiotics and may be used to guide dosing recommendations for ceftobiprole in children. This study is an open-label (all patients will know the identity of the drug) single-dose, pharmacokinetic study in infants and children =3 months to <18 years of age who are medically stable as judged by the clinical investigator and require therapy with antibiotics. Patients will be given a 2-hour i.v. infusion (given directly into the vein) of 7, 10, or 15 mg/kg ceftobiprole. The study population will be grouped according to the following 4 age groups: =12 to <18 years of age; =6 to <12 years of age; =2 to <6 years of age; and =3 months to <2 years of age. Every attempt will be made to include patients of both sexes in each age group. Safety evaluations will include clinical laboratory tests (hematology, serum chemistry, and urinalysis), pregnancy testing, vital signs, physical examination, monitoring of adverse events, and recording of concomitant medications. Patients will be given a single 2-hour i.v. (given directly into the vein) infusion of ceftobiprole. The total duration of the study is approximately 18 days, including screening and posttreatment.

ELIGIBILITY:
Inclusion Criteria:

* Infants (=3 months to <2 years of age) must have been born at =36 weeks of gestation
* Documented or presumed, or be at risk for, bacterial infection(s) and receiving systemic antibiotic therapy
* Stable medical condition

Exclusion Criteria:

* History of drug allergy or hypersensitivity to ß-lactam antibiotics such as penicillins, cephalosporins, or carbapenems
* History of clinically significant cardiac arrhythmia, cystic fibrosis, chronic lung disease associated with abnormal pulmonary function, acute or chronic arthritis
* History of infection with hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2007-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the pharmacokinetics of ceftobiprole when administered as a single dose of 7, 10, or 15 mg/kg in pediatric patients =3 months to <18 years of age who require therapeutic or prophylactic therapy with systemic antibiotics | The total duration of the study is approximately 18 days, including screening and posttreatment with prescreening, Day 1 and Day 2 post treatment

SECONDARY OUTCOMES:
No Secondary Outcomes | 16d

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.